CLINICAL TRIAL: NCT00928369
Title: Clinical Characteristics of Adnexal Masses in Korean Pediatric and Adolescent Patients Under the Age 21 Years
Brief Title: Clinical Characteristics of Patients Under the Age 21 Years Who Underwent Gynecological Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: DooSeok Choi, Samsung Medical Center
Other Study IDs: 2009-04-053
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2009-06

CONDITIONS: Demographic Findings; Presenting Symptoms on First Hospital Visit; Preoperative Radiologic Findings; Operation Method; Histologic Findings

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Young patients with adnexal lesions may have variable presenting symptoms. In this study, we reviewed the clinical characteristics of young Korean patients who took the operation in university hospital with adnexal lesions over the past 14 years.

DETAILED DESCRIPTION:
The incidence of gynecologic surgery during the pediatric and adolescent period remains low. In this age group, the causes of gynecologic surgery were usually divided into three parts, congenital anomalies, genital traumas, and pathologic lesions of genital tract including uterine bady and cervix, ovaries, fallopian tubes, vagina, and vulva. Among these, adnexal masses generally have been the most common cause of gynecologic surgery in the pediatric and adolescent patients. Adnexal lesions span a spectrum of pathology from functional (non-neoplastic), benign to highly aggressive malignant neoplasms. The actual incidence of adnexal lesions in the young women is unknown; however, of the ovarian neoplasms operated on during childhood or adolescence, 10-30% are malignant. Therefore, early detection and adequate management of adnexal lesions are prerequisite for the life saving and future preservation of fertility potential. But until now, there have been limited studies regarding the clinical characteristics of patients with adnexal mass during this period, and most studies have been conducted with small numbers of patients. Therefore, more informations regarding the clinical characteristics of patients with adnexal lesions are very important for the early diagnosis and adequate management of the adnexal lesions in children and adolescents.

In this study, we reviewed the clinical characteristics of 494 young Korean patients who took the operation in university hospital with adnexal lesions over the past 14 years.

ELIGIBILITY:
Inclusion Criteria:

Young women up to 20 years of age who took the gynecologic surgery due to adnexal lesions at the department of Obstetrics and Gynecology, Samsung Medical Center, Seoul, Korea from January, 1995 through March, 2009 were included.

Ages: 1 Year to 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The incidence of gynecologic surgery during the pediatric and adolescent period remains low. In this age group, the causes of gynecologic surgery were usually divided into three parts, congenital anomalies, genital traumas, and pathologic lesions of genital tract including uterine bady and cervix, ovaries, fallopian tubes, vagina, and vulva. Among these, adnexal masses generally have been the most common cause of gynecologic surgery in the pediatric and adolescent patients.
Sampling Method: Non-Probability Sample
Enrollment: 494 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: DooSeok Choi, MD, PhD, Principal Investigator — Samsung Medical Center